CLINICAL TRIAL: NCT04679753
Title: Brainsway Deep TMS System for Treatment of Major Depressive Disorder (MDD) Using Intermittent Theta Burst Stimulation (iTBS) Protocol
Brief Title: Brainsway DTMS for Treatment of MDD Using iTBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0001-03
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Major Depressive Disorder
Keywords: intermittent Theta Burst Stimulation; iTBS; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Brainsway Deep TMS with intermittent Theta Burst Stimulation (iTBS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brainsway DTMS with intermittent Theta Burst Stimulation (iTBS) (Active Comparator): Brainsway DTMS with intermittent Theta Burst Stimulation (iTBS)
  Interventions: Device: Brainsway DTMS with intermittent Theta Burst Stimulation (iTBS)
- Brainsway DTMS with High Frequency Stimulation (HF) (Active Comparator): Brainsway DTMS with High Frequency Stimulation (HF)
  Interventions: Device: Brainsway DTMS with High Frequency (HF) Stimulation

INTERVENTIONS:
Device: Brainsway DTMS with intermittent Theta Burst Stimulation (iTBS) — Brainsway DTMS with iTBS
  Arms: Brainsway DTMS with intermittent Theta Burst Stimulation (iTBS)
Device: Brainsway DTMS with High Frequency (HF) Stimulation — Brainsway DTMS with HF
  Arms: Brainsway DTMS with High Frequency Stimulation (HF)

SUMMARY:
The safety and effectiveness of the BrainsWay deep transcranial magnetic stimulation (DTMS) device for the intended use of Major Depressive Disorder (MDD) using the intermittent theta-burst (iTBS) stimulation protocol will be evaluated in a non-inferiority study, comparing the iTBS treatment with the FDA cleared, (510(k) No. K122288) Brainsway DTMS device to the High Frequency (HF) protocol using the same device.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and efficacy of Brainsway Deep TMS for the treatment of Major Depressive Disorder using the iTBS stimulation protocol, by comparing it to clinical data collected in the Brainsway randomized, controlled Multicenter study (CTP-001-00), using the HF DTMS stimulation protocol used in support of the Brainsway DTMS device 510(k) K122288.

In the post-marketing study, patients will be treated with an intermittent theta burst (iTBS) protocol, using the same Brainsway DTMS device with the same H1-Coil. Furthermore, the treatment paradigm is the same, consisting of TMS sessions performed daily for 5 weeks (20 DTMS sessions). The iTBS stimulation protocol consists of bursts of 3 pulses at 50 Hz, 5 Hz bursts frequency, 2s on and 8s off, 600 pulses per session. The HF stimulation protocol was delivered at 18 Hz, 120% stimulation intensity of the resting MT, 55 trains of 2s duration, inter-train interval (ITI) of 20s, for 1980 pulses per session.

The clinical study design includes multiple measurements of safety and effectiveness parameters.

The primary outcome measure is the change from baseline in HDRS-21 scores at the 5 week visit (after 20 treatment sessions). The success criteria of the study is a non-inferiority margin of 3.0 points.

The secondary efficacy endpoints of the study include evaluation of the response and remission rates, based on HDRS-21 scores, at the 5 week visit, change in CGI-S score from baseline to 6 weeks and response and remission rates based on CGI-S scores at the 6 week visit.

Safety will be assessed at each treatment visit. Patients will be asked to report any adverse event since their previous visit.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Diagnosis of Major Depression Disorder

Exclusion Criteria:

* Other significant Axis I psychiatric disorder with greater impairment than MDD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the change from baseline in HDRS-21 scores at the 5 week visit. | 5 weeks
  Hamilton Depression Rating Scale (HDRS-21 items), where minimum score is 0 and maximum score is 53, and where higher scores mean a worse outcome. The success criteria of the study was a non-inferiority margin of 3.0 points.

SECONDARY OUTCOMES:
HDRS-21 Response and Remission rates | 5 weeks
  Evaluation of the response and remission rates based on HDRS-21 scores
Change in CGI-S score from baseline at the 6 week visit | 6 weeks
  Clinical Global Improvement - Severity Scale (CGI-S), where minimum score is 1 and maximum score is 7, and where higher scores mean a worse outcome.
CGI-S Response and Remission rates | 6 weeks
  Evaluation of the response and remission rates based on CGI-S scores

CONTACTS AND LOCATIONS:
Overall Officials: Oluremi Adefolarin, MD, Principal Investigator — SynapseTMS
Locations (1):
- SynapseTMS, Yorkton, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No